CLINICAL TRIAL: NCT02779790
Title: Effect of Liquid Meal Replacements on Cardiometabolic Risk Factors: A Series of Systematic Reviews and Meta-analyses of Randomized Controlled Trials
Brief Title: Meta-analyses of the Effect of Liquid Meal Replacements on Cardiometabolic Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other); Canadian Diabetes Association (Other); Banting & Best Diabetes Centre (Other)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CIHR-LMRs 2016
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Overweight; Obesity; Type 2 Diabetes
Keywords: Systematic Review and Meta-Analysis; Evidence-Based Medicine; Evidence-Based Nutrition; Clinical Practice Guidelines; Liquid Meal Replacements; Body Weight; Systolic Blood Pressure; Diastolic Blood Pressure; Fasting Blood Glucose; Fasting Blood Insulin; HbA1c; Total Cholesterol; Triglycerides; LDL-C; HDL-C; Controlled Feeding Trials
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Liquid Meal Replacements — An intervention that contains a mixture of protein, carbohydrate, and fat, along with added vitamins and minerals in liquid ready-to-drink or powder formulas that require mixing.
  Other Names: Meal Replacement Shakes

SUMMARY:
Obesity is a major risk factor for cardiovascular disease and diabetes. Weight loss is an important therapeutic goal for overweight and obese patients to reduce their risk of developing cardiovascular disease and diabetes. Liquid meal replacements (LMRs) are simple tools that may aid in weight loss and may improve weight-related risk cardiometabolic risk factors. There is a need to synthesize the evidence on LMRs and cardiometabolic risk to inform clinical practice guidelines. The authors propose to conduct a series of systematic review and meta-analysis of randomized controlled trials to evaluate the effect of LMRs on 4 areas of cardiometabolic risk: markers of adipsoity, glycemic control, established lipid targets, and blood pressure.

DETAILED DESCRIPTION:
Background: Liquid meal replacements (LMRs) provide a mixture of carbohydrate, fat and protein, along with added vitamins and minerals in liquid ready-to-drink form or powder formulas that require mixing. They are designed to mimic a low-calorie meal and serve as a quick and easy source of calories to consume. Behavioral strategy tools are important to assist obese individuals in losing weight and maintaining weight loss. There is evidence that LMRs contribute to weight loss and may reduce related cardiometabolic risk factors.

Need for proposed research: An earlier meta-analysis demonstrated that partial meal replacement plans produced significant weight loss and improved weight-related cardiometabolic risk factors. Several controlled trials have since investigated the effect of liquid meal replacements on body weight and weight-related risk factors for disease. There is a need to update of the evidence of the effect of LMRs on cardiometabolic risk to inform dietary guidelines and public health policy development.

Objective: To synthesize the evidence of randomized controlled trials of the effect of LMRs on body weight, blood pressure, glycemic control and established lipid targets.

Design: The systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by manual searches.

Study selection: The investigators will include randomized controlled trials of >= 2-weeks duration that assess the effect of LMRs versus control diets on body weight, blood pressure, markers of glycemic control and lipid profile.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data.

Outcomes: Four sets of outcomes will be assessed: (1) Markers of adiposity (body weight, BMI, body fat, waist circumference), (2) glycemic control (HbA1c, fasting glucose, and fasting insulin), (3) Established therapeutic lipid targets (LDL-cholesterol, non-HDL-cholesterol, apolipoprotein B, HDL-cholesterol, triglycerides), and (4) blood pressure (systolic blood pressure and diastolic blood pressure).

Data synthesis: Pooled analyses of the mean difference will be performed using the generic inverse variance method. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity because they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will be used only if there are less than 5 included trials. Crossover trials will be assessed via paired analyses. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are >= 10 trials, the study investigators will conduct apriori subgroup analyses by liquid meal replacement type (diabetes-specific formula, soy-based formula and fiber-containing formula), age, health status (presence/absence of type 2 diabetes), comparator, dose, baseline measurements, study design (parallel, crossover), follow-up (<= 3 months, > 3 months) and risk of bias. Meta-regression analyses will assess the significance of categorical and continuous subgroup analyses. When >= 10 trials are available, publication bias will be investigated by funnel plots and formal testing using Egger and Begg tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition and obesity. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed research will synthesize the highest quality evidence from randomized trials and aid in knowledge translation of the effect of LMRs on body weight and related cardiometabolic disease risk. It will strengthen the evidence-base for guidelines, improve health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Trials in humans
* Liquid meal replacement intervention
* Presence of a comparator diet (control diet)
* Diet duration >=2 weeks
* Viable outcome data

Exclusion Criteria:

* Non-human trials
* Observational studies
* Lack of suitable comparator diet
* No viable outcome data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Overweight/Obese, both children and adults.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Markers of adiposity - body weight | Up to 20 years
  Body weight
Markers of adiposity - Body Mass Index | Up to 20 years
  Body Mass Index (BMI)
Markers of adiposity - body fat | Up to 20 years
  Body fat
Markers of adiposity - waist circumference | Up to 20 years
  Waist circumference
Glycemic control - HbA1c | Up to 20 years
  HbA1c
Glycemic control - fasting glucose | Up to 20 years
  fasting glucose
Glycemic control - fasting insulin | Up to 20 years
  fasting insulin
Established therapeutic lipid targets - LDL-cholesterol | Up to 20 years
  LDL-cholesterol (LDL-C)
Established therapeutic lipid targets - apolipoprotein B | Up to 20 years
  Apolipoprotein B (apo B)
Established therapeutic lipid targets - non-HDL-cholesterol | Up to 20 years
  non-HDL-cholesterol (non-HDL-C)
Established therapeutic lipid targets - HDL-cholesterol | Up to 20 years
  HDL-cholesterol (HDL-C)
Established therapeutic lipid targets - triglycerides | Up to 20 years
  Triglycerides
Blood pressure - systolic blood pressure | Up to 20 years
  Systolic blood pressure
Blood pressure - diastolic blood pressure | Up to 20 years
  Diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, MD, PhD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397